CLINICAL TRIAL: NCT04325230
Title: Prognostic Value of Arterial Spin Labeling Brain Perfusion MRI in Term Neonates With Hypoxic-ischemic Encephalopathy
Acronym: BBASL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2020/01
Record Dates: First submitted 2020-03-16; First posted 2020-03-27 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Neonatal Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic-ischemic encephalopathy; Neonate; Perfusion; MRI; Arterial Spin Labeling
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arterial Spin Labeling sequence (Experimental): ASL sequence added to the usual care brain MRI
  Interventions: Device: Arterial Spin Labeling sequence

INTERVENTIONS:
Device: Arterial Spin Labeling sequence — ASL sequence added to the usual care brain MRI

SUMMARY:
The main purpose of this study will be to evaluate the prognostic value at 3 months of life of brain perfusion MRI determined by Arterial Spin Labeling technique in the first week of life of term newborns with hypoxic-ischemic encephalopathy requiring management in neonatal intensive care unit.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy is the result of birth asphyxia due to transitory cerebral blood flow drop during perinatal period. It is the leading cause of neonatal encephalopathy, and thus a major cause of perinatal mortality, morbidity and adverse neurodevelopmental outcome. Usual care brain MRI is critically important in the diagnosis and prognosis. Lasting about 30 to 40 minutes, MRI exam includes successive sequences providing complementary information but none relatively to brain perfusion. Perfusion MRI without contrast media injection is possible using Arterial Spin Labeling (ASL) sequence. ASL is highly suitable for neonates, noninvasiveness, and lasts only 5 minutes. However, only one study assessed ASL as a prognostic factor. The purpose of the study is therefore to perform ASL sequence within usual care brain MRI.

ELIGIBILITY:
Inclusion Criteria:

* neonates with a term ≥ 36 weeks of amenorrhea and birth weight ≥ 1800 g.
* presenting with perinatal asphyxia defined as combination of:

  * an acute perinatal event (such as placental abruption, cord prolapse, and/or severe foetal heart rate abnormalities);
  * and at least one of the following criteria:

    * Apgar score ≤ 5 at 10 minutes of life,
    * mask ventilation or intubation at 10 minutes of life,
    * metabolic acidosis defined as pH < 7 or base deficit ≥ 16 mmol/L or lactates ≥ 11 mmol/L within the first 60 minutes of life on cord or other arterial venous or capillary blood sample.
* patient treated or not with therapeutic hypothermia for 72 hours.
* affiliated patient or beneficiary of a social security scheme.
* informed and signed parental consent.

Exclusion Criteria:

* perinatal arterial ischemic stroke.
* congenital neuro-metabolic disorder.
* severe malformative abnormalities.
* MRI contra-indication.
* Poor understanding of the holders of parental authority

Ages: 1 Day to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcome | 3 months of life (Month 3)
  judged as favorable, or as adverse in case of death or cerebral palsy

SECONDARY OUTCOMES:
Clinical outcome | Month 6, Month 12
  judged as favorable or as adverse
Prognostic performances of ASL | Baseline
  Prognostic performances of ASL in comparison with routinely used MRI parameters
Quality of ASL sequences | Baseline
  according to visual analysis of artifacts and number of negative voxels
Inter-observer agreement of the interpretation of the perfusion data | Baseline
  Intra Class correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No